CLINICAL TRIAL: NCT05258630
Title: Diabetes Homeless Medication Support Randomized Pilot Treatment Development Trial (D-Homes)
Brief Title: Diabetes Homeless Medication Support
Acronym: D-HOMES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2021-317; K23DK118117 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2; Housing Problems; Psychological Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study team will use 1 to 1 allocation to intervention vs. comparison arms. They will stratify based on more and less stable housing in the 12 mo. prior to enrollment.
Who Masked: Outcomes Assessor
Masking Description: Study staff completing post-treatment assessments will be blinded to study condition allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-Homes intervention (Experimental): Behavioral treatments by a diabetes wellness coach as defined below.
  Interventions: Behavioral: Diabetes Homeless Medication Support (D-Homes); Behavioral: Enhanced usual care
- Enhanced usual care (Active Comparator): Brief diabetes educational session by a diabetes wellness coach.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Diabetes Homeless Medication Support (D-Homes) — There will be 10 sessions offered within 12 weeks to participants. Sessions will last approximately 30 minutes. During sessions a diabetes wellness coach will use behavioral activation and motivational interviewing to get to know participants and set goals to improve diabetes care. The coach will encourage a focus on medication adherence behaviors to the extent that participants are willing. The coach will also help with resource and care coordination. The coach will also provide a tailored tool to the patient's needs/goals and tailored diabetes education as needed.
  Arms: D-Homes intervention
Behavioral: Enhanced usual care — Trained diabetes wellness coaches will provide an approximately 15 minutes of instruction about the basic concepts of diabetes. They will use handouts aligned with American Diabetes Association guidelines. They will read these with participants and answer basic questions. Handouts will cover (1) general diabetes knowledge, (2) healthy eating with diabetes, (3) physical activity with diabetes. The coach will also provide a general tool to support medication adherence (e.g. pillbox).

SUMMARY:
This randomized pilot trial of the Diabetes Homeless Medication Support intervention vs. brief diabetes education will test the perception and feasibility of anticipated study procedures and refine randomization and blinding.

DETAILED DESCRIPTION:
This study has an overall goal to develop and pilot test a collaborative care intervention using motivational interviewing and behavioral activation alongside education and psychosocial support to improve medication adherence tailored to the experiences of people experiencing homelessness and diabetes (DH). The investigators' central hypothesis is that medication adherence and diabetes self-care (and eventual glycemic control, health care use/cost) will improve with an intervention tailored to the unique context of DH.

This study will involve addition of a randomization schema to compare D-Homes to brief diabetes education. The study team will enroll participants (n=54), and refine procedures for the randomized trial outcome measures. This includes an assessment of sustained impact of the program at 24-weeks post-treatment. These will complement 12-week post-treatment primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 yrs. or older
2. English-speaking
3. Homelessness by federal definition (HEARTH ACT) in the past 24 mos.
4. Self-reported diagnosis of type 2 diabetes with A1c >7.5%, later verified in medical record and study point-of-care lab test.
5. Plan to stay in local area or be reachable by phone for the next 24 weeks
6. Willingness to work on medication adherence and diabetes self-care

Exclusion Criteria:

1. Inability to provide informed consent (e.g., presence of a legal guardian, prisoners)
2. Active psychosis or intoxication precluding ability to give informed consent
3. Pregnant or lactating people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Vickery, MD, MSc, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin Healthcare, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
As this work is pilot data to inform treatment development for later efficacy testing, we will not share individual participant data. The study team will submit for publication an overall paper describing our results and how they informed future intervention development.

REFERENCES:
- [Derived] Vickery KD, Gelberg L, Hyson AR, Strother E, Carter J, Oranday Perez O, Franco M, Kavistan S, Gust S, Adair E, Anderson-Campbell A, Brito L, Butler A, Robinson T, Connett J, Evans MD, Emmons KM, Comulada WS, Busch AM. Pilot trial results of D-HOMES: a behavioral-activation based intervention for diabetes medication adherence and psychological wellness among people who have been homeless. Front Psychiatry. 2024 Feb 29;15:1329138. doi: 10.3389/fpsyt.2024.1329138. eCollection 2024. PMID 38487573

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | D-Homes Intervention | Enhanced Usual Care
Started | 19 | 19
Completed | 18 | 16
Not Completed | 1 | 3
Not completed — Protocol Deviation w/o increased risk to pt | 1 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Data from one participant from the intervention group and one participant from the enhanced usual care group were not analyzed due to their withdrawal from the study as a result of a protocol deviation.
Groups:
- Total: Total of all reporting groups
Arm/Group | D-Homes Intervention | Enhanced Usual Care | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (10.2) | 51.9 (10.8) | 52.06 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 12 | 26
  White | 0 | 2 | 2
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Experience During the Intervention
Description: The acceptability of the intervention to participants will be measured by the Client Satisfaction Questionnaire, 8-item version, with a score range from 8-32, higher score indicating higher satisfaction.
Time Frame: Assessed at 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | D-Homes Intervention | Enhanced Usual Care
Number analyzed (Participants) | 18 | 18
score on a scale | 29.06 (4.26) | 28.22 (3.66)

2. Primary Outcome: Retention in Assessments
Description: The study team will track enrolled participants who complete both post-treatment assessment visits (12-16 week post-treatment assessment and 24-30 week assessment). Retention will be measured as the percentage of enrolled participants who complete both assessments as assessed at 30 weeks.
Time Frame: Assessed at 30 weeks
Measure: Number; unit: percentage of pts
Arm/Group | D-Homes Intervention | Enhanced Usual Care
Number analyzed (Participants) | 18 | 18
percentage of pts | 100 | 89

3. Secondary Outcome: Change in Glycemic Control
Description: The study team will measure glycemic control using hemoglobin A1c. This will be done on a consistent, validated point-of-care machine using fingerstick blood samples. The study team will compare glycemic control from baseline to 16 weeks and from baseline to 30 weeks.
Time Frame: Assessed at Baseline, 16 weeks, and 30 weeks.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | D-Homes Intervention | Enhanced Usual Care
Number analyzed (Participants) | 18 | 18
percentage of HbA1c
  Baseline | 10.3 (2.1) | 10.4 (2.2)
  16 weeks | 9.7 (2.3) | 9.6 (2.4)
  30 weeks | 9.7 (2.7) | 9.6 (2.4)

4. Secondary Outcome: Psychological Wellness
Description: Psychological wellness is measured with the 5-item Mental Health Inventory (MHI-5), a brief transdiagnostic screening tool attuned to broader concepts of wellbeing and distress than other available measures. MHI-5 scores are computed and transformed on a 0 to 100 point scale with higher scores indicating more wellness. We compare MHI-5 scores from baseline to 16 weeks and from baseline to 30 weeks.
Time Frame: Assessed at baseline, 16 weeks, and 30 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | D-Homes Intervention | Enhanced Usual Care
Number analyzed (Participants) | 18 | 18
score on a scale
  Baseline | 34.4 (24.9) | 39.8 (21.2)
  16 weeks | 38 (20.2) | 37.6 (17.3)
  30 weeks | 34.7 (20.6) | 36.7 (24.4)

5. Secondary Outcome: Diabetes Medication Adherence
Description: As measured by the Adherence to Refills and Medications Scales-Diabetes (ARMS-D), Total scores range from 12-48, with higher values indicating worse outcomes. The study team will compare ARMS-D scores from baseline to 16 weeks and baseline to 30 weeks.
Time Frame: Assessed at Baseline, 16 weeks, and 30 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | D-Homes Intervention | Enhanced Usual Care
Number analyzed (Participants) | 18 | 18
score on a scale
  Baseline | 15.6 (4.6) | 17.2 (3.9)
  16 weeks | 16.0 (5.2) | 16.7 (3.4)
  30 weeks | 15.2 (5.2) | 16.1 (3.7)

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events for the duration of their participation from baseline to 30 weeks for a total of up to 30 weeks.
Arm/Group | D-Homes Intervention | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
Due to the limited resources available in the grant (career development) and delays due to the coronavirus (COVID-19) pandemic, recruitment was closed before reaching our targeted number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT05258630/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05258630/ICF_001.pdf